CLINICAL TRIAL: NCT06504927
Title: Biomarker Discovery in Lung Cancer - Malaysia
Status: Recruiting | Type: Observational
Sponsor: University of Malaya (Other)
Collaborators: MiRXES Pte Ltd (Industry)
Responsible Party: Principal Investigator, Poh Mau Ern, Associate Professor Dr Poh Mau Ern, University of Malaya
Other Study IDs: PRO-MAS-002
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A - High risk cohort: i. Male or female subjects aged 30 and above. ii. No previous history of any cancers. iii. Able to provide X-ray and/or LDCT results. iv. Have one of the following conditions:
  1. COPD
  2. Pulmonary nodules measuring less than 11mm, or deemed not for biopsy by attending physician
  v. Willing to go back for a follow-up X-ray or LDCT scan in the next clinical follow up as per standard of care.
  vi. Willing to provide up to 30mL of blood in month-0 (first visit) and up to 21mL in the next standard of care follow up visit (second visit).
- B - Highly suspicious of lung cancer: i. Male or female subjects aged 30 and above. ii. No previous history of any cancers. iii. Able to provide X-ray and/or LDCT results. iv. Have one of the following conditions:
  1. Suspicious nodules measuring more than 11mm.
  2. Imaging diagnosis suggestive of lung cancer.
  v. Willing to enrol for biopsy for confirmation. vi. Willing to provide up to 39mL of blood in month-0 (first visit) and up to 21mL in the next standard of care follow up visit (second visit).

SUMMARY:
This study aims to

1. Identify biomarkers and signatures to differentiate between high-risk and lung cancer patients.
2. Discover blood-based biomarkers that can be used as an adjunct test to imaging diagnosis to improve patient follow-up.

DETAILED DESCRIPTION:
With existing evidence showing the utility of using liquid biopsy for early cancer detection, the investigators hypothesized that cell-free DNA and/or RNA expression changes during disease progression, and biomarker signature can be derived from the changes in expression levels. The investigators aim to discover and validate RNA and methylated cell-free DNA cancer biomarkers that can discriminate between high-risk and lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 30 and above.
* No previous history of any cancers.
* Able to provide X-ray and/or LDCT results.
* Have either COPD or pulmonary nodules measuring less than 11mm, or deemed not for biopsy by attending physician
* Willing to go back for a follow-up X-ray or LDCT scan in the next clinical follow up as per standard of care.
* Willing to provide up to 30mL of blood in month-0 (first visit) and up to 21mL in the next standard of care follow up visit (second visit).

Exclusion Criteria:

* Subject has received chemotherapy or radiotherapy for cancer treatment, and any other cancer-related treatment.
* Subject is pregnant or lactating (self-declaration).
* Subject is unwilling or unable to provide signed informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort A Subjects in this cohort are recruited if they have either of the following: pre-existing chronic obstructive pulmonary disease (COPD) or are found to have lung nodules smaller than 11mm, or nodules that are deemed not for biopsy by the attending physician.
  Cohort B Subjects in this cohort are highly suspicious of having lung cancer. From the results of the X-ray or LDCT imaging, the subject would have nodules larger than 11mm, or show signs of lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To discover and validate RNA and methylated cell-free DNA cancer biomarkers that can discriminate between high-risk and lung cancer patients. | 3 years
  To discover and validate RNA and methylated cell-free DNA cancer biomarkers that can discriminate between high-risk and lung cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Mau Ern Poh, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT06504927/Prot_000.pdf
  • Informed Consent Form (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT06504927/ICF_002.pdf